CLINICAL TRIAL: NCT05653297
Title: A Randomized Study of The Use of Negative Pressure Wound Therapy in Traumatic Skin & Soft Tissue Loss
Brief Title: Negative Pressure Wound Therapy in Traumatic Skin Loss
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, David Philip Ryad Gadelsayed, Principal Investigator, Assiut University
Other Study IDs: NPWT In Traumatic Wounds
Record Dates: First submitted 2022-11-27; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Post Traumatic Skin Loss
MeSH Terms: interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Group A (Control Group): will undergo conventional dressing daily until the wound is ready for reconstruction, Then coverage of the wound with conventional tie over for 4 days.
- Group B (Experimental Group): NPWT (MEDWAY GROUP VAC) will be applied on a continuous mode between -75 & -150 mm Hg for 4 days per session for indefinite number of sessions until the wound is ready for reconstruction, Then it will be applied after coverage of the wound for 1 session.
  Interventions: Device: Vacuum-Assisted Closure

INTERVENTIONS:
Device: Vacuum-Assisted Closure — NPWT (MEDWAY GROUP VAC) will be applied on post traumatic raw areas until the wound is ready for reconstruction, Then it will be applied over skin graft after coverage
  Groups: Group B (Experimental Group)

SUMMARY:
Assessment of the effectiveness of negative pressure wound therapy on post-traumatic wounds, as regard to :

* The period of granulation tissue formation.
* The infection rate in NPWT in comparison to conventional dressing.
* The rate of graft take after NPWT.
* The length of hospital stay.

DETAILED DESCRIPTION:
Over the last 15 years, negative-pressure wound therapy "NPWT" has become commonly used for treatment of a wide variety of complex wounds. Many clinicians have noted a dramatic response when negative-pressure wound therapy technology has been used, prompting a number of scientific investigations related to its mechanism of action and clinical trials determining its efficacy.

NPWT is a modality that has shown great promise and delivered significantly better results in the clinical care of acute as well as chronic wounds. It is designed to seal the wound site using foam dressing linked to an electronic pump, which applies a pressure ranging from -75 to -150 mmHg. As a matter of fact, NPWT's impact on wound healing appears to be the consequence of multiple effects, each contributing to the overall positive influence on wound healing. Current research indicates that there are four primary NPWT mechanisms of action: Macrodeformation, Microdeformation, Fluid removal and Environmental control of the wound.

Even if the role of NPWT in promoting wound healing has been largely accepted, there is a lack of evidence (few high-level clinical studies) regarding its effectiveness and further research is needed to better understand the mechanisms of action.

Traumatic wounds vary from abrasions and minor skin incisions or tears to wounds with extensive tissue damage or loss and damage to bone and internal organs. Delayed wound healing particularly in difficult wounds is a major concern, It leads to pain, morbidity, prolonged treatment, and require major reconstructive surgery which imposes enormous social and financial burden.

ELIGIBILITY:
Inclusion Criteria:

* No age preference.
* No gender preference.
* Acute traumatic wounds.
* Admitted to the hospital.

Exclusion Criteria:

* Exposed Vessels, Nerves & Organs.
* Active bleeding.
* Ischemic limb.
* Opening into body cavity.
* Vulnerable body organs.
* Necrotic tissue with eschar present.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Post Traumatic Patients with skin & soft tissue loss with no contraindication to use of VAC
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Granulation tissue formation | 2 weeks
  Healthy granulation tissue appears pink to red due to new capillary formation, soft to touch, moist appears "bumpy," and typically painless.
Graft Take | 4 days after coverage
  The graft take assessment by clinical examination

SECONDARY OUTCOMES:
Length of hospital stay | 1 month
  Duration of hospital stay since time of trauma till discharge from hospital after coverage of the wound.

REFERENCES:
- [Background] Orgill DP, Bayer LR. Update on negative-pressure wound therapy. Plast Reconstr Surg. 2011 Jan;127 Suppl 1:105S-115S. doi: 10.1097/PRS.0b013e318200a427. PMID 21200280
- [Background] Bellot GL, Dong X, Lahiri A, Sebastin SJ, Batinic-Haberle I, Pervaiz S, Puhaindran ME. MnSOD is implicated in accelerated wound healing upon Negative Pressure Wound Therapy (NPWT): A case in point for MnSOD mimetics as adjuvants for wound management. Redox Biol. 2019 Jan;20:307-320. doi: 10.1016/j.redox.2018.10.014. Epub 2018 Oct 23. PMID 30390545
- [Background] Peinemann F, Sauerland S. Negative-pressure wound therapy: systematic review of randomized controlled trials. Dtsch Arztebl Int. 2011 Jun;108(22):381-9. doi: 10.3238/arztebl.2011.0381. Epub 2011 Jun 3. PMID 21712971
- [Background] Pappalardo V, Frattini F, Ardita V, Rausei S. Negative Pressure Therapy (NPWT) for Management of Surgical Wounds: Effects on Wound Healing and Analysis of Devices Evolution. Surg Technol Int. 2019 May 15;34:56-67. PMID 31034574
- [Background] El-den S, Reizian A, Yahia A, Zedan A, Shormana M. Effect of Negative Pressure Wound Therapy on Post-traumatic Wound Healing. International Journal of Novel Research in Healthcare and Nursing. 2021;7(3):590-608.
- [Background] Agarwal P, Kukrele R, Sharma D. Vacuum assisted closure (VAC)/negative pressure wound therapy (NPWT) for difficult wounds: A review. J Clin Orthop Trauma. 2019 Sep-Oct;10(5):845-848. doi: 10.1016/j.jcot.2019.06.015. Epub 2019 Jun 20. PMID 31528055